CLINICAL TRIAL: NCT07342140
Title: A Brief and Blended Mindfulness-based Lifestyle Counselling Programme (B-Mindful-Life) for Behavioural Risk Modification Among Caregivers of People With Neurodegenerative Disorders: A Randomised Controlled Trial
Brief Title: Mindfulness-based Lifestyle Modification Programme for Caregivers of People With Neurological Disorders
Acronym: B-Mindful-Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kwok Yan Yan, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23244201
Record Dates: First submitted 2026-01-05; First posted 2026-01-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Caregiver
Keywords: caregivers; behavioral risk; physical activity; mindfulness; ecological momentary; neurological disorders; lifestyle modification; self-care
MeSH Terms: conditions — Motor Activity; Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief and Blended Mindfulness-based Lifestyle counselling programme (B-Mindful-Life) (Experimental): (i) In-Person Mindfulness-based Group Sessions: Two 3-hour group-based session in week 1 and week 5 focused on experiential mindfulness practices. Participants will enhance their self-awareness of positive, neutral, and negative body sensations, feelings, and thoughts while engaging in healthy behaviors, particularly physical activity. (ii) Ecological Momentary Interventions (EMI): Personalized mindfulness-based lifestyle counseling delivered through instant messages, with chat-based support throughout the 8-week intervention period. (iii) Activity Monitoring: All participants will wear an accelerometer-based wristband activity tracker to monitor their physical activity in daily life.
  Interventions: Behavioral: In-Person Mindfulness-based Group Sessions; Behavioral: Ecological Momentary Interventions (EMI); Behavioral: Activity Monitoring
- Brief lifestyle education (Active Comparator): (i) In-person Lifestyle Education Session: A 3-hour group-based session in week 1 focused on general education on lifestyle modification. (ii) Activity Monitoring: All participants will wear an accelerometer-based wristband activity tracker to monitor their physical activity in daily life.
  Interventions: Behavioral: In-person Lifestyle Education Session; Behavioral: Activity Monitoring

INTERVENTIONS:
Behavioral: In-Person Mindfulness-based Group Sessions — The 3-hour group-based session in week 1 focuses on experiential mindfulness practices, and a booster session in week 5 further consolidates these mindfulness techniques, reinforces mindful, healthy lifestyle, and provides peer support. Participants will enhance their self-awareness of positive, neutral, and negative body sensations, feelings, and thoughts while engaging in healthy behaviors, particularly physical activity.
  Arms: Brief and Blended Mindfulness-based Lifestyle counselling programme (B-Mindful-Life)
Behavioral: Ecological Momentary Interventions (EMI) — Participants will receive personalized instant messages with chat-based support throughout the 8-week intervention period. The message content is guided by existing international lifestyle modification guidelines and the Integrated Body-Mind-Spirit Model. The pre-set frequency of regular message delivery is five times per week. The schedule of message delivery will be personalized according to the participants' on-going needs/preferences over the intervention period. Chat-based support will be provided by trained research assistants, who will utilize motivational interviewing techniques to enhance participant compliance and effectiveness.
  Arms: Brief and Blended Mindfulness-based Lifestyle counselling programme (B-Mindful-Life)
Behavioral: In-person Lifestyle Education Session — A 3-hour group-based session in week 1 focused on general education on lifestyle modification based on the HEARTS technical package as recommended by the WHO, and will only receive reminder messages for the two assessment follow-ups. No chat-based support will be provided.
  Arms: Brief lifestyle education
Behavioral: Activity Monitoring — All participants will wear an accelerometer-based wristband activity tracker to monitor their physical activity in daily life.

SUMMARY:
Over 80% of caregivers for individuals with neurodegenerative diseases (ND) engage in significant risk behaviors, particularly physical inactivity, which increases the risk of cardiometabolic diseases (CMD) by 30% and reduces life expectancy by 4-8 years. Despite the health benefits of maintaining healthy behaviors, awareness of behavioral risk management among healthcare professionals and the public is low, and research on this topic for ND caregivers is limited. Given that physical activity (PA) is the most prevalent modifiable risk factor, timely intervention is essential.

International guidelines prioritize PA as a key strategy for caregiver health. However, existing PA interventions often struggle with low compliance due to the physical and emotional challenges caregivers face. Mindfulness-based lifestyle modification might help caregivers better manage physical discomfort, stress, and self-limiting beliefs, thereby supporting sustained PA by improving attentional regulation and psychological flexibility.

The World Health Organization advocates for non-communicable disease (NCD) prevention through brief lifestyle interventions, such as ecological momentary interventions (EMI), which use mobile messaging (e.g., WhatsApp) to deliver personalized health content. This method is particularly valuable for caregivers who find it difficult to access traditional services due to their responsibilities.

A pilot RCT was conducted to compare B-Mindful-Life to brief lifestyle education program in Chinese neurodegenerative disease caregivers, demonstrating promising acceptability, engagement, and effect for increasing PA (NCT06583018). Therefore, this full-power randomized clinical trial aims to rigorously examine its effectiveness and broader impact on this underserved population with several advancement: (i) broaden the population into all neurological disorder caregivers to test for the generalizability of the B-Mindful-Life program; (ii) conduct a 12-month follow-up to assess long-term effects of B-Mindful-Life intervention in real-life settings; (iii) modify outcome measures for targeted assessment. The primary outcome will measure the change in accelerometer-determined, 10-minute bout moderate-to-vigorous physical activity (MVPA) over a 7-day period from baseline to post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults who self-identify as the primary co-residing caregivers of ND patients for ≥3 months. ND is defined as any long-term disorder affecting the nervous system, such as stroke, epilepsy, multiple sclerosis, Parkinson's disease, Alzheimer's disease, traumatic brain injury, migraines, amyotrophic lateral sclerosis, and Huntington's disease;
* Experience of at least mild negative emotions, as indicated by DASS-21 score of Depression subscale ≥10, Anxiety subscale ≥8, or Stress subscale ≥15);
* Have a mobile device (e.g., smartphone, tablet, and laptop) with Internet access; and
* Able to read and communicate in Chinese and give written consent.

Exclusion Criteria:

* Self-reported exercise regimen of great than 150 minutes/week of MVPA (according to the American College of Sports Medicine guidelines);
* Have received (within the past 6 months) or are receiving other physical and/or psychosocial interventions;
* Pregnancy or within 6 months of postpartum; and
* Presence of contraindications, such as a current diagnosis of psychiatric illness (according to the DSM IV-TR, DSM-V, or ICD-10) or severe comorbidities (e.g., severe hearing, vision, or cognitive impairment) that might limit full participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Mean change of time spent on 10-minute bout MVPA over a 7-day period | Baseline (T0) and 2 months (T1)
  For caregivers only, measured by the accelerometer-based wristband activity tracker. The data will be considered valid if the participants wear the activity tracker for ≥10 hours/day for ≥5 days over a 7-day period.

SECONDARY OUTCOMES:
Mean change of time spent on 10-minute bout MVPA over a 7-day period | Baseline (T0), 6 months (T2), and 12 months (T3)
  For caregivers only, measured by the accelerometer-based wristband activity tracker. The data will be considered valid if the participants wear the activity tracker for ≥10 hours/day for ≥5 days over a 7-day period
Mean change of time spent on total MVPA over a 7-day period | Baseline (T0), 2 months (T1), 6 months (T2), and 12 months (T3)
  For caregivers only, measured by the accelerometer-based wristband activity tracker. The data will be considered valid if the participants wear the activity tracker for ≥10 hours/day for ≥5 days over a 7-day period.
Mean change of time spent on sporadic MVPA over a 7-day period | Baseline (T0), 2 months (T1), 6 months (T2), and 12 months (T3)
  For caregivers only, measured by the accelerometer-based wristband activity tracker. The data will be considered valid if the participants wear the activity tracker for ≥10 hours/day for ≥5 days over a 7-day period.
Health-related quality of life | Baseline (T0), 2 months (T1), 6 months (T2), and 12 months (T3)
  For both caregivers and care recipients, measured by EuroQol 5-dimension 5-level questionnaire (EQ-5D-5L). The questionnaire comprises two main components: a description of health status across 5 dimensions (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression), and a numeric value representing the overall health status perceived by the respondents (EQ-VAS). Each dimension is rated from 0 (no problems) to 4 (extreme problems). The scores across the 5 dimensions will be transformed into a utility score based on a validated EQ-5D-5L value set for the Chinese population, with a higher utility score indicating a better health state. The EQ-VAS records an individual's self-rated health on a numeric analogue visual scale, ranging from 0 (the worst health) to 100 (the best health).
Self-reported level of physical activity | Baseline (T0), 2 months (T1), 6 months (T2), and 12 months (T3)
  For caregivers only, measured by International Physical Activity Questionnaire - Short Form. Continuous scores will be calculated according to the standard scoring protocol, which transforms various physical activities into metabolic equivalent (MET)-minutes/week. A higher MET-minutes/week indicates a higher level of physical activity Based on the duration of different physical activities and the calculated MET-minutes/week, participants can also be classified into three categories: Low, Moderate, and High levels of physical activity.
Negative emotions | Baseline (T0), 2 months (T1), 6 months (T2), and 12 months (T3)
  For caregivers only, measured by the Chinese DASS-21 using a one-week recall period, which was developed to measure three related and clinically significant negative emotional states of depression, anxiety and stress. Each item is rated on a 0-3 scale (0="Did not apply to me at all" to 3="Applied to me very much or most of the time"). The score of each subscale ranges from 0-42 and the total score ranges from 0-126, with higher score indicating greater self-reported levels of depression, anxiety and stress.
Caregiver burden | Baseline (T0), 2 months (T1), 6 months (T2), and 12 months (T3)
  For caregivers only, measured by the 12-item Zarit Burden Interview - Short Version (ZBI-SV). Each item is rated on a 0-4 scale (0=Never, 4=Very Often). The total score ranges from 0-48. Higher score indicates heavier caregiver burden. Three domains of ZBI-SV perceived role strain, self-criticism, and negative emotion will also be assessed
Caregiving gains | Baseline (T0), 2 months (T1), 6 months (T2), and 12 months (T3)
  For caregivers only, measured by the Chinese Positive Aspects of Caregiving Scale (C-PACS). Each item is rated on 1-5 scale (1= disagree a lot; 5 = agree a lot). The total score ranges from 10-50. Higher score indicates more positive appraisal towards caregiving. In addition, two domains of the C-PACS, namely enriching life and affirming self will be assessed
Mindfulness | Baseline (T0), 2 months (T1), 6 months (T2), and 12 months (T3)
  For caregivers only, measured by the validated Chinese 32-item Multidimensional Assessment of Interoceptive Awareness (MAIA). Each item is rated on a a 0-5 scale (0=never, 5=always). Higher score indicates higher level of mindfulness. In addition, eight domains of the MAIA, namely noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening and trusting will be assessed.
Self-care behaviors | Baseline (T0), 2 months (T1), 6 months (T2), and 12 months (T3)
  For caregivers only, measured by 20-item Self-Care Inventory (SCI). Each item is rated on a 1 to 5 scale (1=Never, 5=Always). 3 domains of the SCI, namely self-care maintenance, self-care monitoring, and self-care management will be assessed. The score of each domain is derived from the raw summative score using the scoring algorithm proposed by the scale developer, which ranges from 0 to 100. A higher score on the SCI indicates better engagement in self-care in the corresponding domain.
Self-care efficacy | Baseline (T0), 2 months (T1), 6 months (T2), and 12 months (T3)
  For caregivers only, measured by the 10-item Self-Care Self-Efficacy Scale (SCSES). Each item is rated on a 1 to 5 scale (1=No Confident, 5=Extremely Confident). The total score ranges from 10-50. Higher score in SCSES indicates higher level of self-care efficacy.
Attention and meditation levels | Baseline (T0), 2 months (T1), 6 months (T2), and 12 months (T3)
  For caregivers only, measured using a validated electroencephalogram-based headband tracker. Participants will wear the headband with assistance from the outcome assessor before following a standardized audio-guided protocol. Attention and meditation levels will be assessed using a 0-100 rating scale, where a higher score indicates increased focused attention and meditation status, respectively.
Support care needs | Baseline (T0), 2 months (T1), 6 months (T2), and 12 months (T3)
  For care recipients only, measured by the 10-item Palliative care Outcome Scale (POS). The 10 items assess physical symptoms, emotional, psychosocial and spiritual needs, provision of information and practical concerns. Each item is rated on a 0 - 4 scale (0=No burden, 4=Overwhelming problems). The total score ranges from 0-40. Higher score indicates greater unmet support care needs.

OTHER OUTCOMES:
Participant experience of the intervention | 6-month (T2)
  For the experimental group participants, a semi-structured individual interview will be conducted to explore their experiences and identify facilitators and barriers to the implementation and acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jojo Yan Yan Kwok, BNurs, MPH, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, LKS Faculty of Medicine, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data supporting the findings of this study are available upon request from the principal investigator, Prof. Kwok. These data are not publicly available, as they contain information that could compromise the privacy of research participants.